CLINICAL TRIAL: NCT02612285
Title: A Single Arm Study of SNX-5422 in Subjects With TP53 Null Cancers
Brief Title: Study of SNX-5422 in TP53 Null Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment very slow - study could not be enrolled
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN2-010
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open-label administration of SNX-5422 capsules to total 100 mg/m2 every other day for 21 days (total = 11 doses), followed by a 7-day drug-free period. Each treatment cycle will be 28 days. Subjects will repeat this 28-day schedule until the cancer progresses or the subject is unable to tolerate SNX-5422.
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Capsule(s) dosed every other day for 21 days (total 11 doses) out of a 28-day treatment cycle

SUMMARY:
SNX-5422 is a pro-drug of SNX-2112, a potent, highly selective, small-molecule inhibitor of the molecular chaperone heat shock protein 90 (Hsp90). Initial in vitro evidence supports that SNX-5422 may be active against TP53 null tumors irrespective of tumor type .

DETAILED DESCRIPTION:
The tumor suppressor gene TP53 codes for a central regulator of the DNA-damage-response pathway, and its activation leads to cell-cycle arrest and DNA repair, apoptosis, or senescence through both transcription-dependent and transcriptional-independent activities. Somatic TP53 gene alterations are frequent in most human cancers.

SNX-5422 is a pro-drug of SNX-2112, a potent, highly selective, small-molecule inhibitor of the molecular chaperone heat shock protein 90 (Hsp90). Inhibitors of the chaperone protein Hsp90 are of current interest because of the central role that Hsp90 plays in the maturation and maintenance of numerous proteins that are critical for tumor cell viability and growth.

SNX-2112 retains activity in cell lines with loss of the TP53 gene from one of the alleles. SNX-2112 displays good activity in cell lines with TP53 null/TP53 wild type (e.g., MEC-1 [chronic lymphocytic leukemia]) and TP53 null/TP53 mutation (e.g., EBC-1, NCI-H520 [all NSCLC - squamous cell carcinoma]). Even in the most extreme case in which TP53 is lost from both alleles, i.e., the cancer cell is totally devoid of the TP53 gene (e.g., H1299, KATO III, HL-60, SK-MES-1), SNX-2112 retains activity

It appears that SNX-2112 could be active against both hematological and solid tumors with a TP53 null status.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid or hematological TP53 null type cancer.
* No more than 4 prior lines of systemic anti-cancer therapy.
* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older.
* Karnofsky performance score 60
* Life expectancy of at least 3 months.
* Adequate baseline laboratory assessments
* Recovered from toxicities of previous anticancer therapy to CTCAE Grade ≤ 1 with the exception of alopecia.

Exclusion Criteria:

* Treatment with an investigational agent within 30 days prior to the first dose of SNX-5422 or planning to receive an investigational agent during the study.
* Treatment with other anticancer drugs within 28 days or 5 half-lives of anticancer therapy (whichever is shorter) is prohibited from 30 days prior to the first dose of SNX-5422 and throughout the study.
* Radiation treatment within 2 weeks.
* The need for treatment with medications with clinically relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422 (Appendix B).
* Appropriately corrected screening ECG QTc interval 470 msec for females, 450 msec for males.
* Currently receiving medications known to cause QT prolongation AND corrected QTc of 450 msec for females, 430 msec for males.
* Patients with chronic diarrhea of grade 2 or greater despite maximal medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption, including gastric bypass.
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* Seropositive for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Clinically significant glaucoma, retinitis pigmentosa, or macular degeneration.
* Other serious concurrent illness or medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Augusta University, Augusta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - Gabrail Cancer Center Research, Canton, Ohio
  - Wexner Medical Center, Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNX-5422
Started | 1
Completed | 0 (Subject did not complete Cycle 1; no data points recorded)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | SNX-5422
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: Effect of SNX-5422 on tumor progression. Complete remissions plus partial remissions plus stable disease at ≥6 months) will be listed by subject. Tumor measurements made using Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or appropriate hematological malignancy criteria.
Time Frame: 6 months
Population: Subject withdrew from study before any data points gathered
Arm/Group | SNX-5422
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Subject withdrew prior to receiving study drug. No data collected
Description: Subject withdrew prior to receiving study drug. No data collected
Arm/Group | SNX-5422
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No